CLINICAL TRIAL: NCT06175754
Title: Treatment of Reticular Leg Veins: a Prospective, Randomized, Comparative Clinical Trial of a 1064 Nm Nd:YAG Long Pulse Laser, Combined Treatment of a 1064 Nm Nd:YAG Long Pulse Laser and Sclerotherapy Vs. Sclerotherapy Alone.
Brief Title: Laser Treatment of Reticular Leg Veins Vs. Sclerotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Derzhavin Tambov State University (Other)
Responsible Party: Principal Investigator, Oksana Bukina, Director, Clinical Research, Derzhavin Tambov State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DerzhavinTambovSU
Record Dates: First submitted 2023-10-07; First posted 2023-12-19 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-12

CONDITIONS: Reticular Leg Veins
Keywords: reticular veins; long-pulsed Nd:YAG laser; sclerotherapy
MeSH Terms: interventions — Laser Therapy; Lasers; Sclerotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Laser (Active Comparator): to take photo of problem area in the patient's standing position in the room with artificial lighting using the Canon SX510 HS from a distance of 50 cm.
  to measure the maximum diameter of telangiectasia using the Ultrasound Mindray M7 .
  to treat the reticular vein by the Nd:YAG laser with a wavelength of 1064 nm, a 7 mm spot, pulse length of 50 msec and fluency 140 J/cm2
  Interventions: Procedure: Laser ablation
- Laser with Sclerotherapy (Active Comparator): to take photo of problem area in the patient's standing position in the room with artificial lighting using the Canon SX510 HS from a distance of 50 cm.
  to measure the maximum diameter of telangiectasia using the Ultrasound Mindray M7 .
  to treat the reticular vein by the Nd:YAG laser with a wavelength of 1064 nm, a 7 mm spot, pulse length of 15 msec and fluency 70 J/cm2 to inject the 0.3% foam polidocanol with a 5 ml luer-lock syringe through 30 G needle into reticular vein until the vessel disappears.
  Interventions: Procedure: Laser with Sclerotherapy
- Sclerotherapy (Active Comparator): to take photo of problem area in the patient's standing position in the room with artificial lighting using the Canon SX510 HS from a distance of 50 cm.
  to measure the maximum diameter of telangiectasia using the Ultrasound Mindray M7 .
  to inject the 0.5% foam polidocanol with a 5 ml luer-lock syringe through 30 G needle into reticular vein until the vessel disappears.
  Interventions: Procedure: Sclerotherapy

INTERVENTIONS:
Procedure: Laser ablation — Examination, photographing, inclusion in the study, signing of informed consent, randomization, diameter measurement, laser
  Arms: Laser
Procedure: Laser with Sclerotherapy — Examination, photographing, inclusion in the study, signing of informed consent, randomization, diameter measurement, laser plus sclerotherapy
  Arms: Laser with Sclerotherapy
Procedure: Sclerotherapy — Examination, photographing, inclusion in the study, signing of informed consent, randomization, diameter measurement, sclerotherapy
  Arms: Sclerotherapy

SUMMARY:
Treatment of reticular veins with a 1064 nm long-pulsed Nd:YAG laser and combination of a 1064 nm Nd:YAG long pulse laser and sclerotherapy should be no less effective than sclerotherapy alone, and have a frequency of adverse events less then sclerotherapy alone.

DETAILED DESCRIPTION:
Reticular leg veins are mostly an aesthetic problem. Sclerotherapy is considered the gold standard for treatment them. However, this method has a high frequency of long persistent hyperpigmentation which decreases the patients' satisfaction. It is a reason to find another method of treatment. Another possible technique to treat reticular veins is the Nd:YAG long pulse 1064 nm transdermal laser or Nd:YAG laser combined with injection sclerotherapy. There are a few studies comparing sclerotherapy with laser treatment and combined treatment with sclerotherapy. But there are no prospective, randomized, comparative clinical trials of all three methods: the 1064 nm Nd:YAG long pulse laser, combined treatment of a 1064 nm Nd:YAG long pulse laser with sclerotherapy and sclerotherapy alone. The aim of current study is the efficacy assessment of the 1064 nm long-pulsed Nd:YAG laser, combined treatment of the 1064 nm Nd:YAG long pulse laser with sclerotherapy and sclerotherapy alone for the treatment of reticular leg veins and analysis of side effects to establish advantages and disadvantage of these methods and find the best option for treatment of reticular leg veins.

ELIGIBILITY:
Inclusion Criteria:

* women over 18
* reticular veins
* signed informed consent to participate in the study

Exclusion Criteria:

* diabetes mellitus
* pregnancy or lactation
* malignant neoplasms
* inability or unwillingness of the patient to wear compression stockings
* hypersensitivity to the polidocanol, cold, sunlight
* concomitant diseases: bronchial asthma, severe liver and kidney disease, acute thrombosis and thrombophlebitis, infection of the skin and/or soft tissues, infectious diseases, arteriosclerosis, diabetic angiopathy, heart defects requiring surgery, fever, toxic hyperthyroidism, obesity, tuberculosis, sepsis, violation of the cellular composition of the blood, all diseases requiring bed rest, heart disease with decompensation phenomena,
* known hereditary thrombophilia.
* period after treatment of alcoholism
* reception of oral contraceptives
* sedentary lifestyle

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-07-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Disappearance of the reticular vein | 6 months
  The clearing of the vessels on the six-point scale (from 0 to 5 points): 5 - total disappearance of the matting (100% efficacy), 4 - disappearance of around 80%, 3 - disappearance of around 60%, 2 - disappearance of around 40%, 1 - disappearance of around 20%, 0 - no changes.

SECONDARY OUTCOMES:
Pain during the procedure: Numerical Rating Scale | immediately after the procedure
  Estimate of the pain on Numerical Rating Scale. Numerical Rating Scale [NRS] is a measure of pain intensity from 0 to 10 points.
Patient Satisfaction After Treatment | 6 months
  Assessment of patient satisfaction on the 3-point scale :
  no result (0 points), incomplete satisfaction (1 point), complete satisfaction (2 points)
Intensity of hyperpigmentation | 6 months
  Assessment of Intensity of hyperpigmentation on Skin Hyperpigmentation Index (SHI)

CONTACTS AND LOCATIONS:
Overall Officials: Oksana V Bukina, PhD, Principal Investigator — Derzhavin Tambov State University
Locations (1):
- Bukina Oksana Vasilyevna, Tambov, Russia

IPD SHARING:
Plan to Share IPD: Yes
The study data are available to all investigators in the chronic vein disease registry
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From 09 October 2023 to 09 December 2024
Access Criteria: RRT_CVD 1.015
URL: https://www.venousregistry.org/index.php?f=1&id=107

REFERENCES:
- [Background] Nyamekye IK. European Society for Vascular Surgery (ESVS) 2022 clinical practice guidelines on the management of chronic venous disease of the lower limbs. J Med Vasc. 2022 Apr;47(2):53-55. doi: 10.1016/j.jdmv.2022.04.003. Epub 2022 May 23. No abstract available. PMID 35691663
- [Background] Georgiev M. Postsclerotherapy hyperpigmentations: a one-year follow-up. J Dermatol Surg Oncol. 1990 Jul;16(7):608-10. doi: 10.1111/j.1524-4725.1990.tb00088.x. PMID 2362024
- [Background] Goldman MP, Sadick NS, Weiss RA. Cutaneous necrosis, telangiectatic matting, and hyperpigmentation following sclerotherapy. Etiology, prevention, and treatment. Dermatol Surg. 1995 Jan;21(1):19-29; quiz 31-2. doi: 10.1111/j.1524-4725.1995.tb00107.x. PMID 7600016
- [Background] Parlar B, Blazek C, Cazzaniga S, Naldi L, Kloetgen HW, Borradori L, Buettiker U. Treatment of lower extremity telangiectasias in women by foam sclerotherapy vs. Nd:YAG laser: a prospective, comparative, randomized, open-label trial. J Eur Acad Dermatol Venereol. 2015 Mar;29(3):549-54. doi: 10.1111/jdv.12627. Epub 2014 Jul 28. PMID 25069999
- [Background] Ianosi G, Ianosi S, Calbureanu-Popescu MX, Tutunaru C, Calina D, Neagoe D. Comparative study in leg telangiectasias treatment with Nd:YAG laser and sclerotherapy. Exp Ther Med. 2019 Feb;17(2):1106-1112. doi: 10.3892/etm.2018.6985. Epub 2018 Nov 16. PMID 30679981
- [Background] Ozden MG, Bahcivan M, Aydin F, Senturk N, Bek Y, Canturk T, Turanli AY. Clinical comparison of potassium-titanyl-phosphate (KTP) versus neodymium:YAG (Nd:YAG) laser treatment for lower extremity telangiectases. J Dermatolog Treat. 2011 Jun;22(3):162-6. doi: 10.3109/09546631003649679. Epub 2010 Jul 28. PMID 20666669
- [Background] Rogachefsky AS, Silapunt S, Goldberg DJ. Nd:YAG laser (1064 nm) irradiation for lower extremity telangiectases and small reticular veins: efficacy as measured by vessel color and size. Dermatol Surg. 2002 Mar;28(3):220-3. doi: 10.1046/j.1524-4725.2002.01141.x. PMID 11896772
- [Background] Sadick NS. Laser treatment with a 1064-nm laser for lower extremity class I-III veins employing variable spots and pulse width parameters. Dermatol Surg. 2003 Sep;29(9):916-9. doi: 10.1046/j.1524-4725.2003.29250.x. PMID 12930332
- [Background] Moreno-Moraga J, Smarandache A, Pascu ML, Royo J, Trelles MA. 1064 nm Nd:YAG long pulse laser after polidocanol microfoam injection dramatically improves the result of leg vein treatment: a randomized controlled trial on 517 legs with a three-year follow-up. Phlebology. 2014 Dec;29(10):658-66. doi: 10.1177/0268355513502786. Epub 2013 Aug 29. PMID 23989971
- [Background] Fonseca MM, Mocelin FJ, Grill MH, Gianesini S, Miyake K, Argenta R, Pereira AH. Nd:Yag laser combined with injection sclerotherapy in the treatment of reticular veins and telangiectasias (CLaCS method): A triple-blind randomized clinical trial comparing two sclerosing agents associated with same laser patterns. Phlebology. 2023 Apr;38(3):165-171. doi: 10.1177/02683555231153533. Epub 2023 Jan 19. PMID 36657386